CLINICAL TRIAL: NCT03486743
Title: Assessment of Cultural Acceptability of Long Acting Contraception in a Diverse, Urban Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeannette E. South-Paul, Andrew W. Mathieson UPMC Professor and Chair, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Merck IIS# 55000 phase II
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Contraception Behavior
Keywords: LARC contraception cultural acceptance
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: different sites of participant recruitment will be randomized between the use of an informational video during the survey process and no video. The primary focus of the study is the survey that is designed to collect information about cultural perspectives on LARC in the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in the intervention arm will be asked to watch a short educational video on LARC (Long acting reversible contraceptive) and to complete a survey before and after watching the video.
  Interventions: Behavioral: Educational video on LARC
- Control arm (No Intervention): Participants in the intervention arm will only be asked to complete a survey.

INTERVENTIONS:
Behavioral: Educational video on LARC — Participants will watch a short educational video on long acting reversible contraceptive or LARC
  Arms: Intervention arm

SUMMARY:
Preliminary data from our work with teen mothers suggest that many women would benefit from contraception but do not actually make visits nor initiate conversations regarding contraception unless the subject is raised by the clinician. Those coming for primary care visits discuss their conditions and care with family and friends, spreading health care information. A substantial proportion of citizens obtain their health information from friends, family, internet, social media and other non-clinicians. Thus, educating women, even when not coming expressly for contraceptive services, increases more accurate health information throughout their communities and actually identifies fertility needs, ultimately increasing use of contraception.

DETAILED DESCRIPTION:
Seven clinical family medicine health centers will be included in the study. Target participants are women aged 18-45 years old. These clinical sites are community-based health centers within the University of Pittsburgh Medical Center (UPMC) system in greater Pittsburgh that serve as teaching sites for medical, pharmacy and social work students enrolled at the University of Pittsburgh and/or UPMC Family Medicine or clinical pharmacy residents. In 2015, these sites served nearly 32,000 patients of whom more than 60% are women. More than 10,000 females were in the target age group of 18-45 years old and more than half were from underrepresented minority groups. The patients served by these family health centers are diverse across race and ethnicity, family income level, neighborhoods and literacy level . All are managed and documented in the EpicCare electronic medical record system.

We target women aged 18-45 years because this study is designed to assess cultural beliefs regarding Long Acting Reversible Contraception (LARC) in women in general and not specifically those who are seeking contraception. Preliminary data from our work with teen mothers suggest that many women would benefit from contraception but do not actually make visits nor initiate conversations regarding contraception unless the subject is raised by the clinician. Those coming for primary care visits discuss their conditions and care with family and friends, spreading health care information. A substantial proportion of citizens obtain their health information from friends, family, and other non-clinicians. Thus, educating women, even when not coming expressly for contraceptive services, increases more accurate health information throughout their communities and actually identifies fertility needs, ultimately increasing use of contraception.

Seven clinical sites (UPMC Family Health Centers) will be included in the study. The best and low-cost recruitment strategy will be to reach women aged 18-45 years who attend our health centers for womens' health services. Our project team will engage personnel in these health centers and inform them about the proposed study. We will place postcards at the check-in desk, and encourage target women to take a postcards and follow up with the research team if they are interested in participating.

Participants of the project will be identified by the nurses performing initial intakes of patients presenting for care - also called "rooming" the patient. Research assistants will also try to approach patients in the waiting room in the case they were not able to approach them in the examination rooms. Those recruited from each site will be stratified to one of two groups - one for those identifying contraception as the focus of their physician visit and the other group for those seeking other women's health services at the physician visit.

In an effort to improve recruitment, we will work with the clinical staff to understand particular hours during which potential participants are likely to present to the clinic. Flyers will be placed in all seven health centers, In addition, a research assistant will be on site at projected high utilization times. The research assistants will provide information on the study to clinical staff, and will be available to distribute study postcards and answer questions from potential participants. Interested young women will meet with the research assistants for eligibility determination, completion of Institutional Review Board (IRB) consents, and enrollment in the study. Incentives will be provided to all participants enrolled in the study.

Three health centers received a substantial volume of the female patients who were in the specific age group being targeted in the study will be invited to comprise the intervention arm. The rest of the health centers will form the control arm.

It is important that the survey questions reflect the target population's perspectives of using LARC or any contraceptive devices. Both the demographic and cultural surveys will be distributed to women, 18-45 years of age, seeking womens' health services in participating family health centers who expressed interest in the study. Surveys will be completed on a tablet provided by a research assistant or on the participant's own mobile device or personal computer. Participants will be given the option to complete the surveys at the family health center or elsewhere at another time. Women participating in the focus groups are ineligible for participation in the survey.

Participants in the intervention arm will complete both the demographic and the cultural survey. After participating in the survey, the participants in the intervention arm will be asked to watch an educational video on LARC to be taped by a professional team in the Center for Instructional Development & Distance Education (CIDDE) at the University of Pittsburgh. In this video, a family physician skilled in contraceptive education will provide useful and easily understandable information on LARC. The video will include, but is not limited to, the following key topics:

* What types of LARC are available?
* How each LARC method works?
* How and where the LARC method is inserted?
* How long LARC works?
* What are the risks and benefits of each LARC method?
* Can LARC be removed at any time, how it is removed and are there any potential side effects such as slow return of fertility?

A short survey will be distributed to all participants who watched the video in the intervention arm. The survey will include questions on LARC that were similar to the questions included in the survey before watching the video. We will then evaluate both surveys before and after watching the video. The participants will be given the option to complete all study activities at the family health center or elsewhere at another time.

With improved understanding regarding how LARC is perceived through data obtained from the cultural assessment, more targeted education for both clinicians, clinical staff, and patients of childbearing age is possible. Therefore, if the cultural assessment (via focus group feedback and/or survey responses) reveals that patients fear permanent sterilization or believe use of LARC violates religious mores, patient education can be modified to address their specific concerns. These study results may lead to further investigation to change approaches to the target population and allow us to provide better clinical care

Following (1) assessment of historical data on LARC use in the seven health centers prior to this study; (2) perceptions elicited from the focus groups(from phase one of the study); (3) results of the group completing both demographic and cultural surveys; and (4) results of the group completing demographic and cultural surveys and watching the informational video, the final step involves assessing changes in LARC use. Electronic medical records and billing data from the seven health centers will be reviewed to determine LARC utilization across the targeted population served by these health centers and the impact of the interventions on LARC usage.

ELIGIBILITY:
Inclusion Criteria:

* Between age of 18 and 45
* Not currently pregnant
* Did not participate in phase I of the study

Exclusion Criteria:

* Below 18 years or above 45
* Currently pregnant
* Participated in Phase I of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We target women aged 18-45 years because this study is designed to assess cultural beliefs regarding LARC in women in general and not specifically those who are seeking contraception.
Enrollment: 437 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Determine cultural factors that affect women choosing their contraception. | 2 years
  Racial and ethnic minority women are less likely to use LARC than majority women. No studies have primarily focused on contraceptive cultural beliefs of older teens and young women. Potential factors influencing the low LARC usage among teens are inadequate education regarding safety of these methods, misconceptions among clinicians regarding safety of LARC in teens, fewer than ideal numbers of clinicians trained to insert these devices, barriers to obtaining reimbursement for LARC in hospital settings postpartum

SECONDARY OUTCOMES:
Changes in LARC uptake among women seeking contraception. | 2 years
  A variety of myths regarding LARC have been described. Patient myths and misconceptions include that Intra Uterine Devices (IUDs) cause abortions, pelvic inflammatory disease, ectopic pregnancies, weight gain, hair loss, and cancer, among others. Multiple factors affect women in choosing contraception. Each of these potential factors exists in parallel to and may be influenced by the patient's culture (as defined by age, race, ethnicity, religion, family, nationality, language, education, socioeconomic status, and disability.
Studying the effects of using contraception educational video on rates of different contraception methods. | 2 years
  Educating patients about contraception in general, and LARC in specific,is very crucial. In this study we will ask participants to watch a short educational video on LARC and complete a survey before and after the video. This will enable us to understand how educating patients and providing them with information about contraception might affect their perspectives on LARC.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette E. South-Paul, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Latterman Family Health Center, McKeesport, Pennsylvania
  - New Kensington Family Health Center, New Kensington, Pennsylvania
  - UPMC Matilda Theiss Health Center, Pittsburgh, Pennsylvania
  - Squirrel Hill Family Practice, Pittsburgh, Pennsylvania
  - UPMC Bloomfiled-Garfield FHC, Pittsburgh, Pennsylvania
  - Lawrenceville Family Health Center, Pittsburgh, Pennsylvania
  - Shadyside Family Health Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mestad R, Secura G, Allsworth JE, Madden T, Zhao Q, Peipert JF. Acceptance of long-acting reversible contraceptive methods by adolescent participants in the Contraceptive CHOICE Project. Contraception. 2011 Nov;84(5):493-8. doi: 10.1016/j.contraception.2011.03.001. Epub 2011 Apr 27. PMID 22018123
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] Romero L, Pazol K, Warner L, Gavin L, Moskosky S, Besera G, Loyola Briceno AC, Jatlaoui T, Barfield W; Centers for Disease Control and Prevention (CDC). Vital signs: trends in use of long-acting reversible contraception among teens aged 15-19 years seeking contraceptive services-United States, 2005-2013. MMWR Morb Mortal Wkly Rep. 2015 Apr 10;64(13):363-9. PMID 25856258
- [Background] Harper CC, Blum M, de Bocanegra HT, Darney PD, Speidel JJ, Policar M, Drey EA. Challenges in translating evidence to practice: the provision of intrauterine contraception. Obstet Gynecol. 2008 Jun;111(6):1359-69. doi: 10.1097/AOG.0b013e318173fd83. PMID 18515520
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Whitaker AK, Sisco KM, Tomlinson AN, Dude AM, Martins SL. Use of the intrauterine device among adolescent and young adult women in the United States from 2002 to 2010. J Adolesc Health. 2013 Sep;53(3):401-6. doi: 10.1016/j.jadohealth.2013.04.011. Epub 2013 Jun 12. PMID 23763968
- [Background] Damle LF, Gohari AC, McEvoy AK, Desale SY, Gomez-Lobo V. Early initiation of postpartum contraception: does it decrease rapid repeat pregnancy in adolescents? J Pediatr Adolesc Gynecol. 2015 Feb;28(1):57-62. doi: 10.1016/j.jpag.2014.04.005. Epub 2014 May 5. PMID 25555302
- [Background] Okpo E, Allerton L, Brechin S. 'But you can't reverse a hysterectomy!' Perceptions of long acting reversible contraception (LARC) among young women aged 16-24 years: a qualitative study. Public Health. 2014 Oct;128(10):934-9. doi: 10.1016/j.puhe.2014.08.012. Epub 2014 Oct 22. PMID 25369357
- [Background] Greenberg KB, Makino KK, Coles MS. Factors associated with provision of long-acting reversible contraception among adolescent health care providers. J Adolesc Health. 2013 Mar;52(3):372-4. doi: 10.1016/j.jadohealth.2012.11.003. PMID 23427785
- [Background] Rubin SE, Davis K, McKee MD. New york city physicians' views of providing long-acting reversible contraception to adolescents. Ann Fam Med. 2013 Mar-Apr;11(2):130-6. doi: 10.1370/afm.1450. PMID 23508599
- [Background] Russo JA, Miller E, Gold MA. Myths and misconceptions about long-acting reversible contraception (LARC). J Adolesc Health. 2013 Apr;52(4 Suppl):S14-21. doi: 10.1016/j.jadohealth.2013.02.003. PMID 23535052
- [Background] Roncancio AM, Ward KK, Berenson AB. The use of effective contraception among young Hispanic women: the role of acculturation. J Pediatr Adolesc Gynecol. 2012 Feb;25(1):35-8. doi: 10.1016/j.jpag.2011.08.008. Epub 2011 Nov 3. PMID 22051784
- [Background] Doescher MP, Saver BG, Franks P, Fiscella K. Racial and ethnic disparities in perceptions of physician style and trust. Arch Fam Med. 2000 Nov-Dec;9(10):1156-63. doi: 10.1001/archfami.9.10.1156. PMID 11115223
- [Background] Kissling E, Valenciano M, Larrauri A, Oroszi B, Cohen JM, Nunes B, Pitigoi D, Rizzo C, Rebolledo J, Paradowska-Stankiewicz I, Jimenez-Jorge S, Horvath JK, Daviaud I, Guiomar R, Necula G, Bella A, O'Donnell J, Gluchowska M, Ciancio BC, Nicoll A, Moren A. Low and decreasing vaccine effectiveness against influenza A(H3) in 2011/12 among vaccination target groups in Europe: results from the I-MOVE multicentre case-control study. Euro Surveill. 2013 Jan 31;18(5):20390. doi: 10.2807/ese.18.05.20390-en. PMID 23399425
- [Result] deBorja L, Lin C, Maier J, South-Paul JE, Lewis E. Assessment of Cultural Acceptability of Long-Acting Reversible Contraception in a Diverse, Urban Population: Phase II of a Two Phase Study.North American Primary Care Research Group Annual Meeting - NOV 2018 / Chicago, IL (https://www.napcrg.org/conferences/46/sessions/23230)
- [Result] deBorja L. The Role of Social Influence and Usage of Long-Acting Reversible Contraception: Analysis of Survey Responses. North American Primary Care Research Group Annual Meeting - Toronto, ON / NOV. 2019. (https://www.napcrg.org/conferences/2001/sessions/794)
- [Derived] Lin CJ, Maier J, Nwankwo C, Burley C, deBorja L, Aaraj YA, Lewis E, Rhem M, Nowalk MP, South-Paul J. Awareness and Use of Contraceptive Methods and Perceptions of Long-Acting Reversible Contraception Among White and Non-White Women. J Womens Health (Larchmt). 2021 Sep;30(9):1313-1320. doi: 10.1089/jwh.2020.8642. Epub 2020 Dec 9. PMID 33297819